CLINICAL TRIAL: NCT00068172
Title: A Phase I/II Study of PI-88 in Advanced Malignancies (Phase I), and in Advanced Melanoma (Phase II)
Brief Title: Study of PI-88 in Patients With Advanced Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cellxpert Biotechnology Corp. (Industry)
Collaborators: Medigen Biotechnology Corporation (Industry)
Responsible Party: Liz Wilson Director Clinical Operations, Progen Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR88201; PR88201A
Record Dates: First submitted 2003-09-09; First posted 2003-09-10 (Estimated); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — phosphomannopentaose sulfate

INTERVENTIONS:
Drug: PI-88

SUMMARY:
The purpose of this study is to determine whether PI-88 is safe and effective in the treatment of advanced melanoma.

DETAILED DESCRIPTION:
PI-88 is an investigational drug that works by a novel mechanism which may reduce the rate of growth of tumors, and also the spread of cancer cells around the body. It also has an effect upon blood clotting. The purpose of this study is to assess if PI-88 has any benefit to patients with advanced melanoma, as well as to gain further information on the safety of the drug. All patients in the study will receive the study drug at the same dose level. The dose of PI-88 that will be given is based on the dose that was found to be the best in the phase I portion of this study. The drug will be injected subcutaneously (under the skin) once daily for 4 days every week. Patients will be treated with PI-88 for up to 6 months, but if the drug is well tolerated and effective, patients may be offered further treatment with the drug.

ELIGIBILITY:
Inclusion Criteria

* Current diagnosis of metastatic melanoma, where other effective therapy is not available or has failed.
* Measurable disease. Metastatic lesions must be measurable by MRI or CT, and cutaneous lesions by physical examination.
* Aged at least 18 years.
* Have voluntarily given written informed consent to participate in this study.
* Performance status: ECOG 0 - 2 (Karnofsky 70 -100%)
* Life expectancy of at least 3 months.
* Neutrophil count greater than 1.5 x 109/L (1,500/mm3)
* Calculated creatinine clearance, using the Cockcroft-Gault formula, greater than 60 mL/min. If just below 60 mL/min, then GFR greater than 60 mL/min as determined by EDTA or DTPA scan.
* Platelet count at least 100 x 109/L (100,000/mm3)
* Bilirubin less than 1.5 x ULN
* AST and ALT up to 2 x ULN, except in the presence of liver metastases; up to 5 x ULN.
* Prothrombin time less than 1.5 x ULN
* APTT normal (20 - 34 sec)

Exclusion Criteria:

* History of allergy and/or hypersensitivity to anti-coagulants/thrombolytic agents, especially heparin.
* Chemotherapy, investigational or hormonal therapy in the previous 4 weeks.
* Radiotherapy to a major bone marrow bearing area such as pelvis, femoral heads, lumbar-sacral spine, within the previous 4 weeks. Radiotherapy to other sites within the past 2 weeks.
* Uncontrolled infection or serious infection within the past 4 weeks.
* Clinically significant non-malignant disease.
* Known HIV infection or AIDS-related illness.
* Myocardial infarction, stroke or congestive heart failure within the past 3 months.
* Current symptomatic central nervous system involvement, or active brain or meningeal metastases.
* Pregnancy, breast feeding, or women of childbearing potential in whom pregnancy cannot be excluded.
* History of abuse of alcohol, drugs, or other substances.
* History of acute or chronic gastrointestinal bleeding within the last two years, inflammatory bowel disease, any other abnormal bleeding tendency, or patients at risk of bleeding due to open wounds or planned surgery.
* Concomitant use of aspirin (more than 100 mg/day), non-steroidal anti-inflammatory drugs (except COX-2 Inhibitors), heparin, low molecular weight heparin or warfarin (more than 1 mg/day) is ongoing or anticipated during the study period. Low-dose aspirin (up to 100 mg/day) or low-dose warfarin (up to 1 mg/day) is permissible.
* Heparin or low molecular weight heparin within the previous 2 weeks.
* Not recovered from major surgery if conducted prior to the study.
* History of heparin-induced thrombocytopenia, immune mediated thrombocytopenia, thrombotic thrombocytopenic purpura or other platelet disease, or laboratory evidence of anti-heparin antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88
Dates: Start 2001-07; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival by RECIST criteria

SECONDARY OUTCOMES:
Response rate
Time to progression
Overall survival
Biological activity in tumor biopsy specimens

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Health Sciences Center, Aurora, Colorado, United States